CLINICAL TRIAL: NCT02813070
Title: An Open-label Study to Assess Brain Uptake and Safety of Flutemetamol F 18 Injection in Japanese Subjects With Probable Alzheimer's Disease, Subjects With Amnestic Mild Cognitive Impairment and Healthy Volunteers
Brief Title: Comparison of PET Amyloid Imaging in Japanese and Western Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GE067-017
Record Dates: First submitted 2016-06-15; First posted 2016-06-24 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Healthy
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy volunteers (Experimental): 185 MBq [18F] Flutemetamol
  Interventions: Drug: [18F] Flutemetamol
- Mild cognitive impairment (Experimental): 185 MBq [18F] Flutemetamol
  Interventions: Drug: [18F] Flutemetamol
- Alzheimer's Disease (Experimental): 185 MBq [18F] Flutemetamol
  Interventions: Drug: [18F] Flutemetamol

INTERVENTIONS:
Drug: [18F] Flutemetamol — PET brain imaging and Magnetic resonance brain imaging
  Other Names: GE067

SUMMARY:
This was a Phase 2, multicenter study to assess the extent and patterns of [18F] flutemetamol uptake in the brains of 3 groups of Japanese subjects: healthy volunteers (HV), amnestic mild cognitive impairment (aMCI), and probable Alzheimer's disease (pAD), and to assess the reproducibility of brain uptake and of image interpretation. Subjects underwent open-label intravenous (i.v.) administration of Flutemetamol F 18 Injection and Positron emission tomography (PET) imaging of the brain. Blinded visual image reads were performed by 10 independent board-certified readers (5 Japanese and 5 non-Japanese) with nuclear medicine image interpretation experience. The blinded visual assessments were compared with the subject's clinical diagnoses, and the agreement between the image interpretations made by the 2 groups of readers (Japanese and non-Japanese) was determined.

DETAILED DESCRIPTION:
This was a Phase 2, multicenter study to assess the extent and patterns of [18F] flutemetamol uptake in the brains of 3 groups of Japanese subjects: HV, aMCI, and pAD, and to assess the reproducibility of brain uptake and of image interpretation. The 3 comparison groups (HV, aMCI, and pAD) were defined by the subjects' main clinical diagnoses at study entry. Subjects underwent diagnostic quality anatomic brain magnetic resonance imaging (MRI), followed by open-label intravenous (i.v) administration of Flutemetamol F 18 Injection and PET imaging of the brain. Blinded visual image reads were performed by 10 independent board-certified readers (5 Japanese and 5 non-Japanese) with nuclear medicine image interpretation experience. The blinded visual assessments were compared with the subject's clinical diagnoses, and the agreement between the image interpretations made by the 2 groups of readers (Japanese and non-Japanese) was determined. Blinded visual assessments were also compared to quantitative image assessments (standardized uptake value ratio [SUVRs]). Inter-reader and intra-reader agreement was also assessed. Test-retest variability was evaluated following a second administration of Flutemetamol F 18 Injection given to a subset (N=5) of pAD subjects between 1 and 4 weeks after their first administration of Flutemetamol F 18 Injection.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria for all subjects:

1. The subject had at least 6 years of education.
2. The subject was of first-order Japanese descent.
3. The subject exhibited adequate visual, auditory and communication capabilities, and was willing and able to complete standard tests of cognitive function.
4. The subject's general health was adequate to comply with all study procedures, as ascertained by review of their medical history, and laboratory and physical examinations, which was performed within 45 days before the first administration of Flutemetamol F 18 Injection.
5. The subject (and the caregiver, if relevant) was/were compliant and had a high probability of completing the study in the opinion of the investigator.
6. Women were either surgically sterile (had a documented bilateral oophorectomy and/or documented hysterectomy) or were postmenopausal (cessation of menses for more than 2 years).
7. Informed consent was signed and dated by the subject and/or subject's legally acceptable representative, if applicable, in accordance with local regulations.

Inclusion criteria specific for HV:

1. The subject was 25 years or older at the time of obtaining informed consent.
2. The subject had no evidence of cognitive impairment by medical history.
3. The subject had a Mini-Mental State Examination (MMSE) score of =< 27.
4. The subject had a Clinical Dementia Rating (CDR) of 0.
5. The subject had an MRI image as part of the screening visit of sufficient diagnostic quality and consistent with normal brain function (details provided in the associated Imaging Manual) for volume of interest (VOI) definition and partial volume correction.

Inclusion criteria specific for subjects with pAD:

1. The subject was 55 years or older at the time of obtaining informed consent.
2. The subject met National Institute of Neurological and Communicative Disorders and Stroke; Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for clinical pAD and Diagnostic and Statistical Manual of Mental Disorders (DSM-IV]), 4th Edition, criteria for AD (DSM-IV criteria, American Psychiatric Association 1994).
3. The subject had an MMSE score of 15 to 26 (inclusive) and a CDR of 0.5, 1 or 2.
4. The subject had a score of =< 4 on the Modified Hachinski Ischemic scale.
5. The subject had an appropriate caregiver capable of accompanying the subject on all study visits.
6. The subject had an MRI image as part of the screening visit consistent with the diagnosis of pAD and of sufficient diagnostic quality (details provided in the associated Imaging Manual) for VOI definition and partial volume correction.

Inclusion criteria specific for subjects with aMCI:

1. The subject was 55 years or older at the time of obtaining informed consent.
2. The subject met Petersen criteria for aMCI.
3. The subject had an MMSE score of 27 to 30 (inclusive) and a CDR of 0 to 0.5.
4. The subject had a score of =< 4 on the Modified Hachinski Ischemic Scale.
5. The subject had an appropriate caregiver/companion capable of accompanying the subject on all study visits if necessary and applicable according to local regulations.
6. The subject had an MRI image as part of the screening visit consistent with the diagnosis of aMCI and of sufficient diagnostic quality (details provided in Imaging Manual) for VOI definition and partial volume correction.

Exclusion Criteria:

1. The subject was not able to complete the study procedures as judged by the investigator.
2. The subject had received ionizing radiation exposure of more than 1 mSv (except arising from head computed tomography [CT]) in the last 12 months or was determined unsuitable by the investigator as a result of radiation exposure in the past.
3. The subject had a known or suspected hypersensitivity/allergy to [18F] flutemetamol or to any of its excipients.
4. Female subjects who were of childbearing potential, pregnant, or nursing.
5. The subject had a history of alcohol and/or drug abuse within the last 2 years based upon a review of medical records or reported medical history.
6. The subject had a contraindication for MRI or PET (including, but not limited to, claustrophobia, pacemaker, the presence of metallic fragments, or cochlear implant).
7. The subject had participated in a clinical trial using an investigational medicinal product (IMP) within 30 days of dosing.
8. The subject had positive serology for HBs antigen, HCV antibody, HIV antibody or serologic test for syphilis.
9. The subject regularly took medication with a known anticholinergic effect (which could have impaired memory) within the prior 3 months.
10. The subject had a history of head injury associated with significant loss of consciousness that, in the opinion of the investigator, would have interfered with the interpretation of PET images.

Exclusion criteria specific for HV:

1. The subject had any clinically significant medical or neurological condition or any clinically significant abnormality on physical, neurological or laboratory examination.
2. The subject had a family history of pAD (more than 1 first degree relative with the diagnosis of pAD).

Exclusion criteria specific for subjects with pAD and aMCI:

1. The subject had a significant neurological or psychiatric disorder (including, but not limited to, major depression, schizophrenia, mania, etc.) other than pAD that may have affected cognition.
2. The subject had a previous history of clinically evident stroke or significant cerebrovascular disease on brain imaging.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levent Ture, Study Director — GE Healthcare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miki T, Shimada H, Kim JS, Yamamoto Y, Sugino M, Kowa H, Heurling K, Zanette M, Sherwin PF, Senda M. Brain uptake and safety of Flutemetamol F 18 injection in Japanese subjects with probable Alzheimer's disease, subjects with amnestic mild cognitive impairment and healthy volunteers. Ann Nucl Med. 2017 Apr;31(3):260-272. doi: 10.1007/s12149-017-1154-7. Epub 2017 Feb 8. PMID 28181118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 centers in Japan and 1 center in Korea. A total of 87 participants were enrolled and screened in the study, of whom, 17 withdrew prior to dosing and 70 participants received Flutemetamol F 18 injection.
Pre-assignment Details: Participants were assigned into 3 groups based on the baseline diagnosis of probable Alzheimer's disease (pAD), amnestic mild cognitive impairment (aMCI) or healthy volunteers (HVs). All screened participants underwent diagnostic-quality anatomic brain magnetic resonance imaging (MRI) during screening period.
Groups:
- Participants With Probable Alzheimer's Disease: Participants with baseline diagnosis of probable Alzheimer's disease (pAD), received a single intravenous administration of Flutemetamol F 18 injection. Ninety minutes post-injection, participants underwent Positron emission tomography (PET) imaging.
- Participants With Amnestic Mild Cognitive Impairment: Participants with baseline diagnosis of amnestic mild cognitive impairment (aMCI), received a single intravenous administration of Flutemetamol F 18 injection. Ninety minutes post-injection, participants underwent PET imaging.
- Healthy Volunteers: Healthy Volunteers at baseline, received a single intravenous administration of Flutemetamol F 18 injection. Ninety minutes post-injection, participants underwent PET imaging.
Period: Overall Study
Arm/Group | Participants With Probable Alzheimer's Disease | Participants With Amnestic Mild Cognitive Impairment | Healthy Volunteers
Started (Screened participants) | 28 | 23 | 36
Treated (Safety Population) | 25 | 20 | 25
Completed | 25 | 20 | 25
Not Completed | 3 | 3 | 11

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Participants With Probable Alzheimer's Disease: Participants with baseline diagnosis of pAD, received a single intravenous administration of Flutemetamol F 18 injection. Ninety minutes post-injection, participants underwent PET imaging.
- Participants With Amnestic Mild Cognitive Impairment: Participants with baseline diagnosis of aMCI, received a single intravenous administration of Flutemetamol F 18 injection. Ninety minutes post-injection, participants underwent PET imaging.
- Total: Total of all reporting groups
Arm/Group | Participants With Probable Alzheimer's Disease | Participants With Amnestic Mild Cognitive Impairment | Healthy Volunteers | Total
Number analyzed (Participants) | 25 | 20 | 25 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (6.04) | 71.2 (7.28) | 57.4 (9.24) | 67.5 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 11 | 36
  Male | 9 | 11 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Blinded Visual Assessment of Positron Emission Tomography (PET) Imaging and Clinical Diagnosis by Non-Japanese Readers
Description: The performance of Flutemetanol F 18 injection in participants was determined by evaluation of the level of association between the blinded visual assessment of a participant's brain image and the participant's clinical diagnosis by 5 non-Japanese readers, who classified each participant's images as either normal or abnormal (raised) Flutemetanol F 18 uptake.
Time Frame: Up to 90 minutes after investigational medicinal product (IMP) administration
Population: Efficacy population consisted of all participants who had evaluable images following Flutemetamol F 18 injection and evaluable anatomic MRI images. As prospectively planned in the protocol, only participants enrolled with a clinical diagnosis of HV or pAD were included in the analysis of the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Probable Alzheimer's Disease | Healthy Volunteers
Number analyzed (Participants) | 25 | 25
Participants
  Abnormal (positive) participants by Reader A | 23 | 0
  Normal (negative) participants by Reader A | 2 | 25
  Abnormal (positive) participants by Reader B | 23 | 0
  Normal (negative) participants by Reader B | 2 | 25
  Abnormal (positive) participants by Reader C | 23 | 0
  Normal (negative) participants by Reader C | 2 | 25
  Abnormal (positive) participants by Reader D | 23 | 0
  Normal (negative) participants by Reader D | 2 | 25
  Abnormal (positive) participants by Reader E | 23 | 1
  Normal (negative) participants by Reader E | 2 | 24

2. Primary Outcome: Blinded Visual Assessment of Positron Emission Tomography (PET) Imaging and Clinical Diagnosis by Japanese Readers
Description: The performance of Flutemetanol F 18 injection in participants was determined by evaluation of the level of association between the blinded visual assessment of a participant's brain image and the participant's clinical diagnosis by 5 Japanese readers, who classified each participant's images as either normal or abnormal (raised) Flutemetanol F 18 uptake.
Time Frame: Up to 90 minutes after IMP administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Probable Alzheimer's Disease | Healthy Volunteers
Number analyzed (Participants) | 25 | 25
Participants
  Abnormal (positive) participants by Reader F | 23 | 0
  Normal (negative) participants by Reader F | 2 | 25
  Abnormal (positive) participants by Reader G | 22 | 1
  Normal (negative) participants by Reader G | 3 | 24
  Abnormal (positive) participants by Reader H | 23 | 0
  Normal (negative) participants by Reader H | 2 | 25
  Abnormal (positive) participants by Reader I | 23 | 1
  Normal (negative) participants by Reader I | 2 | 24
  Abnormal (positive) participants by Reader J | 23 | 1
  Normal (negative) participants by Reader J | 2 | 24

ADVERSE EVENTS:
Time Frame: The safety of participants was monitored during the course of the study till 24-hours post administration of Flutemetanol F 18 injection.
Description: Analysis was performed on safety population that included all participants who received any dose of Flutemetanol F 18 injection in the study.
Arm/Group | Participants With Probable Alzheimer's Disease | Participants With Amnestic Mild Cognitive Impairment | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.